CLINICAL TRIAL: NCT02210442
Title: Educaguia Project: Clinical Trial, Randomised by Clusters, to Assess the Effectiveness of a Strategy With Educational Games to Implementation pf Clinical Practice Guidelines to Family Medicine Residents in Spain.
Brief Title: Effectiveness of Educational Games to Implementation Clinical Practice Guidelines to Family Medicine Residents in Spain.
Acronym: EDUCAGUIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gerencia de Atención Primaria, Madrid (Other Government)
Collaborators: Fondo de Investigacion Sanitaria (Other)
Responsible Party: Principal Investigator, Isabel Del Cura-Gonzalez, PhD. MD, Gerencia de Atención Primaria, Madrid
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 11/0047
Record Dates: First submitted 2014-04-29; First posted 2014-08-06 (Estimated); Last update posted 2018-02-07 (Actual); Status verified 2018-02

CONDITIONS: Health Knowledge, Attitudes, Practice
Keywords: educational games; clinical practice guideline; family medicine; primary health care; cluster clinical trial
MeSH Terms: conditions — Behavior | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Educaguia intervention (Experimental): Implementation of practice clinical guidelines with educational games
  Interventions: Behavioral: educaguia intervention
- Control group (Active Comparator): Implementation of clinical practice guidelines with standard practice care
  Interventions: Other: control group

INTERVENTIONS:
Behavioral: educaguia intervention — Health professionals (residents) play with educational games in order to acquire knowledge and skill about management of clinical practice guidelines.
  Arms: Educaguia intervention
Other: control group — Health professional will learn how to manage a clinical practice guidelines with standard clinical practice.
  Arms: Control group

SUMMARY:
A multicenter study to evaluate the effectiveness of a teaching strategy based on the incorporation of educational games with simulated settings versus usual practice based on diffusion for the implementation of clinical practice guidelines in Family Medicine Residency Program. The impact of the new strategy will be measured in improving knowledge and skill acquisition in clinical decision making of Family Medicine Residency Program after 6 months. Effectiveness will also be measured a month and 12 months after intervention.

DETAILED DESCRIPTION:
Objective: To evaluate the effectiveness of educational games to implementation practice guidelines to acquire skills in clinical decision-making by family medicine residents in Spain.

Secondary objectives: To describe the strategies utilized in Residency Program in Family Medicine in Spain to teach the use of practice guidelines. To identify barriers and facilitators for the use of practice guidelines for family medicine residents.

Setting: Unit Family Medicine in Spain. Study design: Multicentric cluster randomised controlled clinical trial. Population: Family Medicine Residents of second and third year. Sample size: 394 residents (197 in each arm). The randomization units will be units (clusters). The units of analysis are professionals (residents). Variables: Main outcome variable measured in both groups: assess of skill levels and number of correct answers about clinical questions in diabetes, anxiety disorders, antibiotic prescription and insomnia clinical practice guidelines in primary care.

Sociodemographic variables and educational variables for each subject and variables regarding Residency Program in Family Medicine.

Intervention: EDUCAGUIA plan. Incorporating educational games online for each guideline.

Statistical Analysis: Primary and secondary effectiveness. Adjusting by contextual and individual variables factors with mixed effects models (lineal regression) (dependent variable: points obtained in educational games in each guide).

ELIGIBILITY:
Inclusion Criteria:

* Second and third year residents in Family Medicine Program.

Exclusion Criteria:

* Giving up the Family Medicine Program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2017-01-17 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Assessing clinical decision-making skills | Change from Baseline skills at 6 months
  Outcomes of a test designed to assess problem solving and clinical decision making skills about anxiety disorders, diabetes, insomnia and prescription antibiotics prescription after six months after intervention.

SECONDARY OUTCOMES:
Assessing clinical decision-making skills | Change from Baseline at 1 month and 12 months
  Outcomes of a test designed to assess problem solving and clinical decision making skills about anxiety disorders, diabetes, insomnia and prescription antibiotics prescription after 1 month and 12 months after intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Isabel del Cura, MD PhD, Principal Investigator — Reserch Unit. Gerencia de Atención Primaria Madrid, Servicio Madrileño de Salud. Madrid. Spain.
Locations (1):
- Gerencia de Atención Primaria, Madrid, Spain

REFERENCES:
- [Background] Del Cura-Gonzalez I, Lopez-Rodriguez JA, Sanz-Cuesta T, Rodriguez-Barrientos R, Martin-Fernandez J, Ariza-Cardiel G, Polentinos-Castro E, Roman-Crespo B, Escortell-Mayor E, Rico-Blazquez M, Hernandez-Santiago V, Azcoaga-Lorenzo A, Ojeda-Ruiz E, Gonzalez-Gonzalez AI, Avila-Tomas JF, Barrio-Cortes J, Molero-Garcia JM, Ferrer-Pena R, Tello-Bernabe ME, Trujillo-Martin M; Educaguia Group. Effectiveness of a strategy that uses educational games to implement clinical practice guidelines among Spanish residents of family and community medicine (e-EDUCAGUIA project): a clinical trial by clusters. Implement Sci. 2016 May 17;11:71. doi: 10.1186/s13012-016-0425-3. PMID 27189180
- [Derived] Del Cura-Gonzalez I, Ariza-Cardiel G, Polentinos-Castro E, Lopez-Rodriguez JA, Sanz-Cuesta T, Barrio-Cortes J, Andreu-Ivorra B, Rodriguez-Barrientos R, Avila-Tomas JF, Gallego-Ruiz-de-Elvira E, Lozano-Hernandez C, Martin-Fernandez J; Educaguia Group. Effectiveness of a game-based educational strategy e-EDUCAGUIA for implementing antimicrobial clinical practice guidelines in family medicine residents in Spain: a randomized clinical trial by cluster. BMC Med Educ. 2022 Dec 24;22(1):893. doi: 10.1186/s12909-022-03843-4. PMID 36564769